CLINICAL TRIAL: NCT04450056
Title: Assessing Changes in Breastmilk Composition Over Time Among Pakistani Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Founding Chair, Centre of Excellence in Women and Child Health, Aga Khan University
Other Study IDs: 2020-3676-10314b
Record Dates: First submitted 2020-06-22; First posted 2020-06-29 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Breast Milk Collection; Infant Development
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breastmilk sample Rectal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother-infant pairs: Mothers with a term-born (>37 weeks gestation) infant whom they are exclusively or predominantly breastfeeding at 1 month postpartum. Mothers must be enrolled in the MaPPS Trial (ClinicalTrials.gov Identifier: NCT03287882).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In Pakistan, breastfeeding is widely practiced. National data suggests that 94% of infants <2 years of age receive breastmilk at some point. However, the introduction of complementary foods often occurs early. At 3 months of age, it is suggested that only 54% of Pakistani infants are exclusively breastfed. This declines with each month of age. Because the production and release of breastmilk is influenced by the frequency and intensity of suckling, early initiation of complementary feeding can reduce breastmilk output. Given that complementary foods are introduced early within Pakistan, we hypothesize that breastmilk composition will change between 1 and 3 months postpartum among those mother-infant pairs if nutritive complementary foods are introduced early (i.e., before 6 months). In this study, we aim to better understand how breastmilk composition changes over time among infants recruited at 1 month of age who are exclusively breastfed or receive only non-nutritive feeds. This is a substudy to the Matiari emPowerment and Preconception Supplementation (MaPPS) Trial (ClinicalTrials.gov Identifier: NCT03287882).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the MaPPS Trial
* Mothers must report practicing exclusive or predominant breastfeeding (i.e., breastmilk only or breastmilk and non-nutritive feeds only)
* The infant must be term-born (>37 weeks gestation)
* Infant must be 1 month + 14 days old at the time of recruitment
* Mothers must be willing to provide a complete breastmilk expression from one breast (either via breast pump or hand expression)
* Able to provide informed consent

Exclusion Criteria:

* Mother reports mixed feeding of her infant with nutritive feeds (i.e., any provision of formula or animal milk)
* The infant was born preterm (earlier than 37 weeks gestation)
* Mother does not wish to provide a complete breast expression of one breast

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Mothers and infants enrolled in the MaPPS Trial in Matiari District, Pakistan.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in breastmilk macronutrient composition | 1 and 3 months postpartum
Change in breastmilk micronutrient composition | 1 and 3 months postpartum

SECONDARY OUTCOMES:
Change in breastmilk bioactive composition | 1 and 3 months postpartum
Change in breastmilk microbiome | 1 and 3 months postpartum
Change in infant microbiome | 1 and 3 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Matiari Research and Training Centre, Matiari, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Please contact the Primary Investigator directly for more details.